CLINICAL TRIAL: NCT04425694
Title: Implementation and Evaluation of an Electronic Early Warning Score (e-EWS) System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Lingnan University (Other); Tuen Mun Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: e-EWS 20200526
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: patient safety; electronic Early Warning Score system; human factors
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- F3B ward staff: The e-EWS system will be implemented in a selected surgical ward (F3B ward) in Tuen Mun Hospital. All F3B ward staff will use the system and evaluate its effectiveness.
  Interventions: Device: e-EWS system

INTERVENTIONS:
Device: e-EWS system — The e-EWS system is connected to a physiological monitor, which takes various physiological measurements. The system has an auto-charting module, which automatically captures patients' physiological measurements in an electronic chart (e-chart) and calculates their EWS. All the information in the auto-charting module is then wirelessly transferred to a central display in the ward's nurses station. The central display shows patients' status in terms of EWS and issues alerts when any EWS has exceeded a set threshold. The e-EWS system is not only capable of auto-charting but also provides an alert mechanism to help nurses detect early deterioration.

SUMMARY:
Early Warning Score (EWS) is a tool designed to help clinicians efficiently identify and track patients who have or develop acute illness, and make timely clinical responses. The calculation and charting of EWSs at Tuen Mun Hospital (TMH) is a manual process at present. The purpose of this study is to automate the EWS calculation and charting process using an electronic EWS (e-EWS) system. However, while the e-EWS system could potentially reduce ward staff's workload and improve patient safety, its effectiveness can only be realized through good human factors (HF) design that matches users' expectations, requirements and work practices. Therefore, our aim is to carry out HF methods in order to inform design of the e-EWS system before its implementation in a selected surgical ward in the hospital. After its implementation, we will also conduct evaluation of the e-EWS system to assess its effectiveness with respect to clinical outcomes.

DETAILED DESCRIPTION:
Early Warning Score (EWS), also known as "track-and-trigger" system, is a tool designed to help clinicians efficiently identify and track patients who have or develop acute illness, and make timely clinical responses. An EWS is calculated based on values from a number of physiological parameters (e.g. respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness, and temperature) to obtain an aggregated score, which indicates a patient's health status. It is mostly used by ward nurses to monitor their patients; when a patient's EWS has exceeded a set threshold, the nurse should attend to the patient more closely and consider for intervention e.g. call a doctor. The philosophy of EWS is that it improves patient safety by enabling ward staff to detect patients' deterioration early so that timely intervention can be administered within the "golden period for treatment".

In the U.K., an EWS system called the National Early Warning Score (NEWS) was first released in 2012 (NEWS, 2012). The NEWS was the first system to standardize the calculation and charting of acute-illness severity and has been widely adopted across the National Health Service (NHS). Recently, in December 2017, NEWS2 has been released and it is an updated version of the NEWS (NEWS2, 2017). NEWS2 can be readily computerized and has already been integrated with some NHS hospitals' electronic health record systems. The Updated Report of a Working Party of NEWS2 states that "There are potential advantages of automated calculation of the NEW score and automated alert systems." (p. 6). Therefore, the objective of this proposed study is to implement and evaluate an electronic EWS (e-EWS) system in a selected surgical ward at Tune Mun Hospital (TMH).

At TMH, the current practice of obtaining ward patients' EWS is a manual process: firstly, a care giver measures a patient's specified physiological parameters by using the appropriate monitoring instruments; secondly, the care giver writes down the values of the parameters on a paper chart; thirdly, the paper chart is handed over to a nurse; and finally, the nurse calculates the EWS. The process is performed on a designated regular time interval.

There are two main drawbacks of the manual EWS process: firstly, it is inefficient because there are usually multiple patients in a ward and some physiological variables take time to measure. Therefore, in a busy ward, missed physiological measures and irregular measurement-taking intervals are often reported. These problems lead to staff ignoring EWS calculations. Secondly, when EWS are calculated, nurses often do so for patients who already show deteriorating conditions. This counters the original intent of EWS, which is to help identify patients with early signs of deterioration. These drawbacks compromise clinicians' ability to detect patient deterioration early, which could potentially compromise patient safety.

A potential solution is to automate the manual EWS process. Some hospitals in Hong Kong, for example, Tseung Kwan O Hospital has already adopted an e-EWS system in some of its wards. The e-EWS system is connected to a physiological monitor, which takes various physiological measurements. The system has an auto-charting module, which automatically captures patients' physiological measurements in an electronic chart (e-chart) and calculates their EWS. All the information in the auto-charting module is then wirelessly transferred to a central display in the ward's nurses station. The central display shows patients' status in terms of EWS and issues alerts when any EWS has exceeded a set threshold. The e-EWS system is not only capable of auto-charting but also provides an alert mechanism to help nurses detect early deterioration.

However, while the e-EWS system could potentially reduce ward staff's workload and improve patient safety, its effectiveness can only be realized through good HF design that matches users' expectations, requirements and work practices.

ELIGIBILITY:
Inclusion Criteria:

* All F3B ward nursing staff

Exclusion Criteria:

* Staff not in F3B ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the runner nurses and the ward manager in a selected surgical ward (F3B ward) at Tuen Mun Hospital (TMH).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of successful detection of deteriorating cases | from the beginning of the study to the 6th month later
Changes in the number of cardiopulmonary resuscitations (CPRs) | from the beginning of the study to the 6th month later
Changes in the number of ICU or high dependency unit transfer | from the beginning of the study to the 6th month later
Changes in the number of assistance calls to doctors | from the beginning of the study to the 6th month later

SECONDARY OUTCOMES:
Changes in application-specific self-efficacy | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's perceived usefulness of the e-EWS system | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's perceived ease of use of the e-EWS system | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's perceived behavioral control | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's attitude towards the e-EWS system | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's intention to use | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's perceived work performance | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's perceived workload | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in the quality of patient care | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in the workflow | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in the accuracy of the technology | from the beginning of the study to the 6th month later
  This outcome will be measured by the 7-point Likert scale, with scores ranging from 1 (very strongly disagree) to 7 (very strongly agree).
Changes in ward staff's personal experiences in current clinical unit | from the beginning of the study to the 6th month later
  This outcome will be measured by the 4-point Likert scale, with scores ranging from 1 (strongly disagree) to 4 (strongly agree).
Comments and suggestions of the system | from the beginning of the study to the 6th month later
  Ward staff's opinions will be collected by a semi-structured interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuen Mun Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Royal College of Physicians. National Early Warning Score (NEWS): Standardising the assessment of acute illness severity in the NHS. Report of a working party. London: RCP, 2012.
- [Background] Royal College of Physicians. National Early Warning Score (NEWS) 2: Standardising the assessment of acute-illness severity in the NHS. Updated report of a working party. London: RCP, 2017.
- See also: Nielsen, J. (2012, June 4). How Many Test Users in a Usability Study? — http://www.nngroup.com/articles/how-many-test-users/